CLINICAL TRIAL: NCT01317498
Title: Effect of Routine Viral Load Monitoring on Clinical and Immunological Outcomes and Antiretroviral Drug Resistance on Patients Taking First-line Antiretroviral Drugs in Vietnam
Brief Title: The VMVN Study: Virological Monitoring in Viet Nam
Acronym: VMVN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Bach Mai Hospital (Other); Roche Molecular Systems, Inc (Industry)
Responsible Party: Principal Investigator, Todd Pollack, Assistant Professor in Medicine, Part-time, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010P000334
Record Dates: First submitted 2011-03-09; First posted 2011-03-17 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: HIV Infection; AIDS
Keywords: ART; antiretroviral; treatment; Vietnam; Asia; viral load
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Monitoring (Placebo Comparator): The patients in the standard monitoring arm will receive routine laboratory monitoring as provided to all patients in public HIV clinics in Vietnam, including CD4 count, complete blood count, and liver functions tests every 6 months.
  Interventions: Other: Standard Care
- Virological Monitoring (Active Comparator): The patients in the virological monitoring arm will have routine laboratory monitoring as in the standard monitoring arm and in addition will have a viral load test performed every 6 months while in treatment. The first test will be done 6 months after initiating ART.
  Interventions: Other: Virological Monitoring

INTERVENTIONS:
Other: Standard Care — CD4, liver function and CBC every 6 months
  Arms: Standard Monitoring
Other: Virological Monitoring — Viral Load test every 6 months
  Arms: Virological Monitoring

SUMMARY:
The purpose of the study is to test the hypothesis that the addition of routine viral load testing to the standard laboratory monitoring of HIV patients on first-line antiretroviral treatment (ART) in Vietnam will result in better clinical outcomes for patients.

DETAILED DESCRIPTION:
The optimal strategy for monitoring antiretroviral therapy (ART) in resource-limited settings (RLS) is unknown. In developed countries, routine monitoring with CD4 count and viral load (VL) testing is standard practice. In RLS, however, limitations in the availability of the technology for VL testing, and in financial resources to pay for VL testing, mean that few developing countries provide VL testing as part of the routine monitoring of patients on ART. Instead, ART is monitored primary by clinical examination with CD4 testing where available. This strategy has been endorsed by the most recent WHO guidelines for ART (WHO, 2010).

Standard laboratory monitoring of patients on ART in Vietnam includes CD4 testing every 6 months, where available. In many rural areas of the country, CD4 testing is not available and only clinical monitoring is used.

In this study we will test the hypothesis that routine viral monitoring every 6 months for patients on first-line ART will result in significantly higher rates of virological suppression and decrease the incidence of death or new or recurrent AIDS-defining illnesses by 50% within three years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18
* Confirmed HIV infection
* Not currently taking ART
* Meets Vietnam MOH criteria for ART (THROUGH OCTOBER 2011:CD4<250 cells/mm3, WHO Clinical Stage IV, or WHO clinical stage III with CD4<350 cells/mm3; FROM NOVEMBER 2011: CD4<350 cells/mm3, OR WHO Clinical Stage III or IV)
* Completes required Vietnam MOH ART adherence training
* Signs written informed consent form

Exclusion Criteria:

* Any ART use within the previous 3 months
* History of treatment failure on first-line ART or known resistance to first-line ART.
* Unable or unwilling to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2011-04 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Death or new/recurrent AIDS-Defining (WHO Clinical Stage IV) Illnesses | 3 years
  The number of deaths and/or new/recurrent WHO Clinical Stage IV clinical illnesses that occur over 3 years of follow-up in each group.
Virological Suppression | 3 years
  The percentage of patients in each group who are still on treatment at 3 years who have virological suppression, defined as an HIV viral load below the level of laboratory detection.

SECONDARY OUTCOMES:
Time to identification and diagnosis of treatment failure. | 3 years
  To calculate the difference in times in the 2 groups from the first emergence of active viral replication (defined as a detectable viral load) to identification and diagnosis of treatment failure.
Time from virological treatment failure to switch to second line ART. | 3 years
  We will calculate the mean time from virological treatment failure to switch to second line ART in both groups.
Resistance mutations | 3 years
  The difference in resistance mutation patterns at the diagnosis of virological treatment failure in each group.
Sensitivity and specificity of WHO criteria for treatment failure | 3 years
  To determine the sensitivity and specificity of WHO criteria for treatment failure among patients on first-line ARV in Vietnam.
Cost-benefit analysis | 3 years
  To evaluate and compare the costs and benefits of adding routine VL testing to standard laboratory monitoring for patients on first-line ART in Vietnam. In the event that the trial shows a benefit in the primary outcome of decreased number of deaths plus WHO Stage 4 clinical events, the analysis will evaluate the cost per life saved and the cost per outcome event avoided. The analysis will also include a cost per quality-adjusted life year saved.

CONTACTS AND LOCATIONS:
Overall Officials: Todd M Pollack, MD, Principal Investigator — Beth Israel Deaconess Medical Center; Pham T Thuy, MD, PhD, Principal Investigator — Bach Mai Hospital, Hanoi, Vietnam; Julian Elliott, MBBS, PhD, Principal Investigator — Alfred Hospital, Melbourne, Australia; Donn J Colby, MD, MPH, Principal Investigator — Center for Applied Research on Men and Health
Locations (1):
- Bach Mai Hospital, Hanoi, Vietnam

REFERENCES:
- See also: Harvard Medical School AIDS Initiative in Vietnam — http://www.haivn.org